CLINICAL TRIAL: NCT02604290
Title: Kinesio Taping Method for Chronic Mechanical Low Back Pain: a Randomised Controlled Trial
Brief Title: Kinesio Taping Efficacy in Chronic Low Back Pain Treatment (KITALO)
Acronym: KITALO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Collaborators: Cardenal Herrera University (Other); Hospital Arnau de Vilanova (Other)
Responsible Party: Principal Investigator, Julio Domenech, MD-PhD, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSK063
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Chronic Low Back Pain
Keywords: Kinesio taping; Neuromuscular taping; Targeted treatment; Chronic low back pain; Randomised controlled trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kinesio Taping method (Experimental): The tape is applied depending on the physical examination:
  * Muscular technique is placed along paravertebral muscles if back pain in flexion or extension improves when skin/fascial mobilisation is applied in the direction of paravertebral muscle fibers; the base is placed up or down if the mobilisation direction is up or down respectively.
  * Space technique is placed horizontally over the painful spinal segmental level if back pain in flexion or extension improves when skin/fascial mobilisation is applied approaching to a central point.
  * Fascia technique is placed horizontally over the painful area in paravertebral muscles if back pain in flexion or extension improves when skin/fascial mobilisation is applied transverse to the paravertebral muscle fibers.
  Interventions: Device: Kinesio Taping method
- Kinesio Taping sham (Sham Comparator): The tape is applied with 0% tension, horizontally over two non-tender to palpation spinal segmental levels. The patient is kept in neutral position.
  Interventions: Device: Kinesio Taping sham

INTERVENTIONS:
Device: Kinesio Taping method — The tape is applied depending on the physical examination:
  * Muscular technique is placed along paravertebral muscles if back pain in flexion or extension improves when skin/fascial mobilisation is applied in the direction of paravertebral muscle fibers; the base is placed up or down if the mobilisation direction is up or down respectively.
  * Space technique is placed horizontally over the painful spinal segmental level if back pain in flexion or extension improves when skin/fascial mobilisation is applied approaching to a central point.
  * Fascia technique is placed horizontally over the painful area in paravertebral muscles if back pain in flexion or extension improves when skin/fascial mobilisation is applied transverse to the paravertebral muscle fibers.
  Arms: Kinesio Taping method
Device: Kinesio Taping sham — The tape is applied with 0% tension, horizontally over two non-tender to palpation spinal segmental levels. The patient is kept in neutral position.
  Arms: Kinesio Taping sham

SUMMARY:
The purpose of this study is to determine whether the kinesio taping method is effective in the treatment of chronic (more than six months duration) low back pain.

DETAILED DESCRIPTION:
Hypothesis: Kinesio taping treatment in patients with chronic low back pain, in which fascial mobilisation represents a treatment effect modifier, reduces pain and disability and improves quality of live, in comparison with simulated kinesio taping.

Objective:

* Primary objective: To evaluate kinesio taping method effectiveness at short term (1 month) and medium term (6 months) - pain, disability and quality of live - in patients with chronic low back pain.
* Secondary objective: To analyze the influence of fear-avoidance beliefs, catastrophizing ideas and anxiety-depression presence in kinesio taping method effectiveness for chronic low back pain patients.

Method:

Chronic low back pain patients are recruited from the outpatient rehabilitation service of a health area of Valencia which serves a population of 320,000 inhabitants.

The study has been planned for a difference of 3 points in the Roland Morris questionnaire, as these values have been recognized as clinically relevant . Considering an alpha of 0.05 and beta of 0.9 for comparison of means of two tails , 24 patients per group is the required sample size to detect changes in disability. Considering a loss of 20 % of the participants, the study sample is set to 62 patients.

Addressing the CONSORT guidelines, a flow chart describing the situation during the course of the trial is draw; including all patients invited , the number of those who refuse to participate before randomization , the assignment to each treatment arm, losses during follow-up and possible crosslinking.

Patients who agree to participate in the study are randomly assigned to one of two intervention groups. The allocation was made by a list generated by computer using the Statistical Package for the Social Sciences (SPSS 19), supervised by an statistical outside of the investigator team . Concealment of randomization sequence is maintained with hidden cards in numbered opaque envelopes.

The duration of treatment is 4 weeks , changing the tape with a weekly frequency. Basic rules of postural control and stabilization and the pattern of exercises proposed by the Spanish Society for Rehabilitation and Physical Medicine are given prior to randomization.

The evaluation of results is done through self-administered questionnaires to be completed by the patients ever before clinic visits .

The primary results will be obtained by intention to treat analysis. Descriptive statistics will be obtained expressing continuous variables in mean (standard deviation) or median (quartiles) according to their normal or not, categorical variables in number (percentage) and expressing in all cases the confidence interval of 95%. The normal distribution was checked by Kolmogorov test to determine the use of parametric or non-parametric tests. For comparison of continuous variables between groups the Student t test or the Mann-Whitney test will be used according to the type of distribution. For comparison of categorical variables the chi-square test or Fisher will be used test according to the type of distribution. Changes in intra-group in continued variables at 4 weeks and 6 months will be analyzed with the Student t test for paired samples variables. To assess whether there are differences between the two groups in pain, disability and different variables analysis of covariance (ANCOVA) will be held, one for each dependent variable. In all tests, the independent variable is the group, while the covariate variable will be the baseline for each dependent variable. It will be necessary to have comparable levels in both groups to correctly interpret the results of ANCOVA. Therefore, several Student t tests, one for each dependent variable considering each group as an independent variable in each case, will be made. To assess whether changes in the 2 groups are produced differently, multiple ANOVA analysis for each dependent variable will be performed. In all cases, the independent variable is the group and the time data are collected. This analysis examines only the possible presence of interactions. In addition, correlations between the study variables will be evaluated, using Pearson's r or Rho Spearman according to the type of distribution. Two models of multiple linear regression will be applied with pain and disability as dependent variables and age, sex, pain catastrophizing, fear-avoidance, sick leave, time to progression, anxiety-depression as independent variables.

The project will follow existing in Spain and the European Union guidelines for the protection of patients in clinical trials with respect to collection, storage and custody of personal data.

All eligible patients are given oral and written information ( informed consent) about the study and the two treatment modalities. Specifically they are informed about they can leave the study at any time without giving any explanation and that this decision will not affect the continuation of his regular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Chronic low back pain least 6 months duration.
* Improvement of pain with mobilization of skin/fascias in physical examination.
* Signature of informed consent.

Exclusion Criteria:

* Having had previous treatment experience with kinesio taping method.
* Presence of components of neuropathic pain (radiculopathy, lumbar canal stenosis).
* Specific origin pain (vertebral fracture, tumor or nerve column structures, spondyloarthropathy, spondylodiscitis).
* Prior spine surgery.
* Mental retardation, severe mental illness, substance abuse or dependency, illiteracy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2016-11-14 (Actual)

PRIMARY OUTCOMES:
Change in "Roland Morris Disability Questionnaire" | pretreatment, 4 weeks, 6 month
  Assess activity limitations due to back pain. Consists of 24 statements. Patients were asked to answer yes or no to each statement. Each positive answer is worth one point with scores ranging from 0 (no disability) to 24 (severely disabled). The Spanish version has been validated.

SECONDARY OUTCOMES:
Change in "Fear Avoidance Beliefs Questionnaire" | pretreatment, 4 weeks, 6 month
  measure fear and avoidance beliefs related to low back pain. It consists of 16 sentences related to physical activity (first 5 items) and work (last 11 items). The patient has to rate each sentence from 0 (totally disagree) to 6 (totally agree). The score range is 0 to 96, with a higher value reflecting a higher degree of fear avoidance beliefs. Two subscales are defined. "Factor 1" is composed of items 6, 7, 9, 10, 11, and 12 and reflects fear-avoidance beliefs about work. "Factor 2" is composed of items 2 to 5 and reflects fear-avoidance beliefs about physical activities. The Spanish version has been validated.
Change in "Pain Catastrophizing Scale" | pretreatment, 4 weeks, 6 month
  This scale assess patient negative and exaggerated orientation to painful stimuli. It has 13 item and comprises three dimensions: a) rumination; b) magnification, and c) hopelessness. Each item scores on a 5-point Likert scale (0 not at all 1 a little, 2 moderately, 3 very much, 4 all the time. The score range is 0 to 52, with a higher value reflecting a higher degree of pain catastrophizing. The Spanish version has been validated
Change in "Hospital Anxiety and Depression subscale" | pretreatment, 4 weeks, 6 month
  This scale is used for screening mood and anxiety disorders. Consists of a 7-item anxiety subscale and a 7-item depression subscale. Each item scores on a 4-point Likert scale (0 as much as I always do; 1 not quite so much; 2 definitely not so much; 3 not at all ), giving maximum subscale scores of 21 for depression and anxiety, respectively. The Spanish version has been validated.

OTHER OUTCOMES:
Charlson Comorbidity Index | pretreatment
Adverse effects | 4 weeks
Change in "EuroQol-5D-5L (EuroQol 5 dimensions and 5 levels)" | pretreatment, 4 weeks, 6 month
  This scale is a generic measure of health. Comprises 5 dimensions (mobility, self care, usual activities, pain/discomfort, anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The digits for 5 dimensions can be combined in a 5-digit number describing the respondent's health state.The EuroQol VAS records the respondent's self-rated health on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. The Spanish version is available.
Change in "Numerical Rating Scale" | pretreatment, 4 weeks, 6 month
  Assess pain intensity, involves asking patients to rate the pain from 0 to 10 (an 11-point scale), with the understanding that 0 represents one end of the pain intensity continuum (" no pain") and 10 represents the other extreme of pain intensity (" pain as bad as it could be").

CONTACTS AND LOCATIONS:
Overall Officials: María Lourdes Peñalver Barrios, MD, Principal Investigator — Hospital Arnau de Vilanova, Valencia, Spain; Julio Domenech Fernández, MD, PhD, Study Director — Hospital Arnau de Vilanova, Valencia, Spain; Juan Francisco Lisón Párraga, MD, PhD, Study Director — Cardenal Herrera CEU University
Locations (1):
- Hospital Arnau de Vilanova, Valencia, Spain

REFERENCES:
- [Background] Kent P, Mjosund HL, Petersen DH. Does targeting manual therapy and/or exercise improve patient outcomes in nonspecific low back pain? A systematic review. BMC Med. 2010 Apr 8;8:22. doi: 10.1186/1741-7015-8-22. PMID 20377854
- [Background] Parreira Pdo C, Costa Lda C, Hespanhol LC Jr, Lopes AD, Costa LO. Current evidence does not support the use of Kinesio Taping in clinical practice: a systematic review. J Physiother. 2014 Mar;60(1):31-9. doi: 10.1016/j.jphys.2013.12.008. Epub 2014 Apr 24. PMID 24856938
- [Background] Paoloni M, Bernetti A, Fratocchi G, Mangone M, Parrinello L, Del Pilar Cooper M, Sesto L, Di Sante L, Santilli V. Kinesio Taping applied to lumbar muscles influences clinical and electromyographic characteristics in chronic low back pain patients. Eur J Phys Rehabil Med. 2011 Jun;47(2):237-44. Epub 2011 Mar 24. PMID 21430611
- [Background] Castro-Sanchez AM, Lara-Palomo IC, Mataran-Penarrocha GA, Fernandez-Sanchez M, Sanchez-Labraca N, Arroyo-Morales M. Kinesio Taping reduces disability and pain slightly in chronic non-specific low back pain: a randomised trial. J Physiother. 2012;58(2):89-95. doi: 10.1016/S1836-9553(12)70088-7. PMID 22613238
- [Background] Kachanathu SJ, Alenazi AM, Seif HE, Hafez AR, Alroumim MA. Comparison between Kinesio Taping and a Traditional Physical Therapy Program in Treatment of Nonspecific Low Back Pain. J Phys Ther Sci. 2014 Aug;26(8):1185-8. doi: 10.1589/jpts.26.1185. Epub 2014 Aug 30. PMID 25202177
- [Background] Parreira Pdo C, Costa Lda C, Takahashi R, Hespanhol Junior LC, Luz Junior MA, Silva TM, Costa LO. Kinesio taping to generate skin convolutions is not better than sham taping for people with chronic non-speci fi c low back pain: a randomised trial. J Physiother. 2014 Jun;60(2):90-6. doi: 10.1016/j.jphys.2014.05.003. Epub 2014 Jun 10. PMID 24952836